CLINICAL TRIAL: NCT04264130
Title: Evaluation of the Effect of Artemisinin-based Combination Therapies on Urinary Schistosoma Haematobium When Administered for the Treatment of Malaria Co-infection
Brief Title: Effect of Artemisinin-based Combination Therapies on Schistosomiasis on Malaria Co-infection
Acronym: SACT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre de Recherche Médicale de Lambaréné (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEI-006/2018
Record Dates: First submitted 2020-02-06; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Schistosomiasis Haematobia
MeSH Terms: conditions — Schistosomiasis haematobia | interventions — pyronaridine tetraphosphate, artesunate drug combination; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- artemisinin-based combination therapies (Active Comparator): subjects given Artemisinin-based combined therapies according to the study instruction
  Interventions: Drug: Artesunate-Pyronaridine; Drug: Artemether-Lumefantrine
- non-artemisinin drugs (Sham Comparator): subjects given non artemisinin based combined therapies like describe in the study protocol
  Interventions: Drug: Artefenomel-Ferroquine

INTERVENTIONS:
Drug: Artesunate-Pyronaridine — Subjects received artesunate-pyronaridine according to their body weight once per day for three days.
  Other Names: Pyramax
  Arms: artemisinin-based combination therapies
Drug: Artemether-Lumefantrine — subjects received artemether-lumefantrine according to their body weight twice per day for three days.
  Other Names: Coartem
  Arms: artemisinin-based combination therapies
Drug: Artefenomel-Ferroquine — Subject received a single dose of artefenomel-ferroquine according to their body weight
  Arms: non-artemisinin drugs

SUMMARY:
Open labelled, non randomized study to evaluate the effects of Artemisinin based Combined Therapies(ACTs) on schistosomiasis since Praziquantel (PZQ) which is presently the drug of choice for treating Schistosomiasis (STS), is ineffective on immature stages and there is known parasite resistance. ACTs when combined with PZQ, targeting different stages of the life cycle has shown some effectivity.

DETAILED DESCRIPTION:
Study population included all subjects in study area who signed a written Informed Consent Form diagnosed with Malaria- STS co-infection. Those excluded were treated with PZQ prior 6 weeks, have drug intolerance or pregnant. At Inclusion, Basic Demographic data was recorded and urine samples analysed. During the follow up visits, urine samples were collected on D28 and D42 (6 weeks post treatment). Post treatment assessment was done on urine samples collected on at least two consecutive days and at the end of follow up, all subjects were treated with a single dose pf PZQ (40 mg/kg) as recommended by WHO.

ELIGIBILITY:
Inclusion Criteria:

* Malaria infection diagnosed by Rapid Diagnostic Tests (RDTs) or thick blood smear
* Urinary schistosomiasis diagnosed by presence of Schistosoma haematobium eggs in the urine before malaria treatment
* Written informed consent

Exclusion Criteria:

* Patients treated with PZQ during the previous 6 weeks
* Known intolerance /allergy to any study drug
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Egg Reduction Rate (ERR) | Day 28
  Evaluate ERR conferred by ACTs as treatment of infection with Schistosoma hematobia
Egg Reduction Rate (ERR) | Day 42
  Evaluate ERR conferred by ACTs as treatment of infection with Schistosoma hematobia

SECONDARY OUTCOMES:
Cure Rate (CR) | Day 28
  CR of ACTs on Schistosoma haematobia
Cure Rate (CR) | Day 42
  CR of ACTs on Schistosoma haematobia

CONTACTS AND LOCATIONS:
Overall Officials: Rella Zoleko Manego, Principal Investigator — Centre de Recherches Medicales de Lambarene, Lambarene, Gabon
Locations (1):
- Centre de Recherches Medicales de Lambarene, Lambaréné, Gabon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zoleko-Manego R, Okwu DG, Handrich C, Dimessa-Mbadinga LB, Akinosho MA, Ndzebe-Ndoumba WF, Davi SD, Stelzl D, Veletzky L, Kreidenweiss A, Nordmann T, Adegnika AA, Lell B, Kremsner PG, Ramharter M, Mombo-Ngoma G. Effectiveness of antimalarial drug combinations in treating concomitant urogenital schistosomiasis in malaria patients in Lambarene, Gabon: A non-randomised event-monitoring study. PLoS Negl Trop Dis. 2022 Oct 31;16(10):e0010899. doi: 10.1371/journal.pntd.0010899. eCollection 2022 Oct. PMID 36315579